CLINICAL TRIAL: NCT04685265
Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Oral Doses of anle138b, and to Characterise the Effect of Food of anle138b in Mild to Moderate Parkinson's Disease
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of anle138b in Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MODAG GmbH (Industry)
Collaborators: Aptuit (Industry); Quotient Sciences (Industry); Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: anle138b-P1-02; 2020-004869-38 (EudraCT Number)
Record Dates: First submitted 2020-12-17; First posted 2020-12-28 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease
Keywords: anle138b; alpha-Synuclein; Oligomer modulator; Multiple System Atrophy; Parkinson Disease; Alzheimer Disease; Neurodegenerative diseases; Tauopathies; Amyloid
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body; Multiple System Atrophy; Alzheimer Disease; Neurodegenerative Diseases; Tauopathies | interventions — 3-(1,3-benzodioxol-5-yl)-5-(3-bromophenyl)-1H-pyrazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is double-blind. Treatment assignment will not be known to the subjects, the sponsor or the staff who are involved in the clinical evaluation of the subjects and the analysis of data. The randomisation schedule and disclosure envelopes will be generated by an unblinded statistician at Quotient Sciences.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anle138b (Active Comparator): 150 mg and higher dosage
  Interventions: Drug: anle138b
- Placebo (Placebo Comparator): Matching placebo dosage
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: anle138b — capsule containing excipient and anle138b
  Arms: anle138b
Drug: Placebo — matching placebo capsule containing excipient
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability and blood levels of orally administered anle138b as well as the effect of food and early signs of efficacy in patients with mild to moderate Parkinson´s disease.

DETAILED DESCRIPTION:
This is a two centre, double-blind, randomised, placebo-controlled, multiple ascending dose study in patients with mild to moderate Parkinson´s disease. It is planned to enrol up to 5 cohorts. Cohorts A-C consist of up to 8 subjects. In Cohorts A and B, subjects will be randomly assigned to receive multiple ascending oral doses of anle138b or matching placebo (6 active investigational medicinal product [IMP], 2 placebo per cohort in cohorts A-C) for 7 days in a sequential escalating manner. Subjects in cohort A and B will be dosed once dialy and subjects in cohort C will be dosed twice a day. Subjects in Cohorts A and B will also receive an additional single oral dose of active IMP or matching placebo on Day 9 of the study for an assessment of the effect of food on the PK of anle138b in PD patients. Subjects in cohort D will be randomly assigned to receive QD doses of anle138b or matching placebo (placebo vs 150 mg vs 300 mg; 1:1:1) for 7 days in fasted state. Subjects in Cohort E will be randomly assigned to receive QD doses of either 300 mg anle138b or matching placebo (1:1) for 28 days taken in the non-fasted state.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with a diagnosis of idiopathic PD as defined by the Movement Disorders Society criteria (either fulfilling criteria for "Clinically Established PD" or for "Clinically Probable PD").
* Body mass index (BMI) 18.5 to 35.0 kg/m2 or 18.5 to <40.0 kg/m2 (Cohorts D and E) as measured at screening.
* Hoehn and Yahr stage I-III (able to walk unaided).
* Stable medication for PD for 1 month prior to screening at Quotient and anticipated over the study period.
* No history of dementia.
* Must be willing and able to communicate and participate in the whole study.
* Must provide written informed consent.
* Must agree to adhere to the contraception requirements defined in the study protocol.

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1.
* Subjects who are, or are immediate family members of, a study site or sponsor employee.
* Evidence of current SARS-CoV-2 infection.
* History of any drug or alcohol abuse in the past 2 years.
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type).
* A confirmed positive alcohol breath test at screening or admission.
* Current smokers and those who have smoked within the last 12 months. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission (Cohorts A to C only).
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months (Cohorts A to C only).
* Females of childbearing potential including those who are pregnant or lactating (all female subjects must have a negative highly sensitive serum or urine pregnancy test). A woman is considered of childbearing potential unless she is permanently sterile (hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) or is postmenopausal (had no menses for 12 months without an alternative medical cause and a serum follicle-stimulating hormone [FSH] concentration ≥40 IU/L).
* Male subjects with pregnant or lactating partners.
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening.
* Clinically significant abnormal coagulation (Cohort E only), clinical chemistry, haematology or urinalysis as judged by the investigator.
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results.
* History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or gastrointestinal disease or psychiatric disorder, as judged by the investigator.
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active.
* Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood.
* Subjects who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies other than their regular medication according to the referral letter from NUH, and/or up to 2 g of paracetamol per day and/or HRT, in the 14 days before IMP administration.
* Subjects who are taking, or have taken, in the 14 days before IMP administration the drug warfarin.
* Subjects who are taking, or have taken, in the 14 days before IMP administration any drug that is considered to interfere with the objectives of the study, as determined by the concomitant medication oversight committee.
* Subjects who have participated in Cohorts A to C of this study will not be allowed to participate in Cohorts D or E, and subjects who have participated in Cohort D will not be allowed to participate in Cohort E.
* Failure to satisfy the investigator of fitness to participate for any other reason.
* Subjects who have a new headache with features suggestive of raised intracranial pressure, including papilloedema, vomiting, posture-related headache, or headache on waking from sleep (Cohort E only).
* Subjects who have a new headache with focal neurological symptoms, or non-focal neurological symptoms such as change in personality or memory, or an unexplained headache that becomes progressively severe, or an unexplained headache in anyone previously diagnosed with cancer (Cohort E only).
* Medical history or evidence of mass occupying lesion in brain or spinal cord or history of spinal cord injury, which could preclude the procedure of lumbar puncture and CSF collection (Cohort E only).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events in PD patients with multiple ascending doses of anle138b taken in the fasted state (cohorts A-C + D). | Day 1 to day 14-16: cohorts A-C; day 1 to week 6 post dosing: cohort D
  Adverse events
Incidence of treatment-emergent adverse events in PD patients with multiple ascending doses of anle138b taken in the fed state (Cohorts A and B). | From fed dosing (day 9) to day 12-14
  Adverse events
Incidence of treatment-emergent changes in vital signs in PD patients with multiple ascending doses of anle138b taken in the fasted state (cohorts A-C + D). | Day 1 to week 1 post dosing: cohorts A-C; day 1 to week 6 post dosing: cohort D
  Blood pressure
Incidence of treatment-emergent changes in vital signs in PD patients with multiple ascending doses of anle138b taken in the fasted state (cohorts A-C + D). | Day 1 to week 1 post dosing: cohorts A-C; day 1 to week 6 post dosing: cohort D
  Heart rate
Incidence of treatment-emergent changes in vital signs in PD patients with multiple ascending doses of anle138b taken in the fasted state (cohorts A-C + D). | Day 1 to week 1 post dosing: cohorts A-C; day 1 to week 6 post dosing: cohort D
  Oral temperature
Incidence of treatment-emergent changes in vital signs in PD patients with multiple ascending doses of anle138b taken in the fed state (Cohorts A and B). | From fed dosing to 1 week post dosing
  Blood pressure
Incidence of treatment-emergent changes in vital signs in PD patients with multiple ascending doses of anle138b taken in the fed state (Cohorts A and B). | From fed dosing to 1 week post dosing
  Heart rate
Incidence of treatment-emergent changes in vital signs in PD patients with multiple ascending doses of anle138b taken in the fed state (Cohorts A and B). | From fed dosing to 1 week post dosing
  Oral temperature
Incidence of treatment-emergent ECG changes in PD patients with multiple ascending doses of anle138b taken in the fasted state (cohorts A-C + D). | Day 1 to week 1 post dosing: cohorts A-C; day 1 to week 6 post dosing: cohort D
  Electrocardiogram (ECG) parameters including QT interval corrected for heart rate using Fridericia's formula (QTcF)
Incidence of treatment-emergent ECG changes in PD patients with multiple ascending doses of anle138b taken in the fed state (Cohorts A and B). | From fed dosing to 1 week post dosing
  Electrocardiogram (ECG) parameters including QT interval corrected for heart rate using Fridericia's formula (QTcF)
Incidence of treatment-emergent changes in physical examination in PD patients with multiple ascending doses of anle138b taken in the fasted state (cohorts A-C + D). | Day 1 to week 1 post dosing: cohorts A-C; day 1 to week 6 post dosing: cohort D
  Physical examination findings
Incidence of treatment-emergent changes in physical examination in PD patients with multiple ascending doses of anle138b taken in fed state (Cohorts A and B). | From fed dosing to 1 week post dosing
  Physical examination findings
Incidence of treatment-emergent changes in clinical laboratory parameters in PD patients with multiple ascending doses of anle138b taken in the fasted state (cohorts A-C + D). | Day 1 to day 8
  Clinical laboratory Tests: Hematology
Incidence of treatment-emergent changes in clinical laboratory parameters in PD patients with multiple ascending doses of anle138b taken in the fasted state (cohorts A-C + D). | Day 1 to day 8
  Clinical chemistry: Renal function tests
Incidence of treatment-emergent changes in clinical laboratory parameters in PD patients with multiple ascending doses of anle138b taken in the fasted state (cohorts A-C + D). | Day 1 to day 8
  Clinical chemistry: Hepatic enzymes
Incidence of treatment-emergent changes in clinical laboratory parameters in PD patients with multiple ascending doses of anle138b taken in the fasted state (cohorts A-C + D). | Day 1 to day 8
  Clinical chemistry: Electrolytes
Incidence of treatment-emergent changes in clinical laboratory parameters in PD patients with multiple ascending doses of anle138b taken in the fasted state (cohorts A-C + D). | Day 1 to day 8
  Clinical chemistry: Creatine kinase
Incidence of treatment-emergent changes in clinical laboratory parameters in PD patients with multiple ascending doses of anle138b taken in fed state (Cohorts A and B). | From fed dosing to 24 hours post dosing
  Clinical laboratory Tests: Hematology
Incidence of treatment-emergent changes in clinical laboratory parameters in PD patients with multiple ascending doses of anle138b taken in fed state (Cohorts A and B). | From fed dosing to 24 hours post dosing
  Clinical chemistry: Renal function tests
Incidence of treatment-emergent changes in clinical laboratory parameters in PD patients with multiple ascending doses of anle138b taken in fed state (Cohorts A and B). | From fed dosing to 24 hours post dosing
  Clinical chemistry: Hepatic enzymes
Incidence of treatment-emergent changes in clinical laboratory parameters in PD patients with multiple ascending doses of anle138b taken in fed state (Cohorts A and B). | From fed dosing to 24 hours post dosing
  Clinical chemistry: Electrolytes
Incidence of treatment-emergent changes in clinical laboratory parameters in PD patients with multiple ascending doses of anle138b taken in fed state (Cohorts A and B). | From fed dosing to 24 hours post dosing
  Clinical chemistry: Creatine kinase
Incidence of treatment-emergent adverse events in PD patients with multiple ascending doses of anle138b taken 28 days in the non-fasted state (cohort E). | Day 1 to week 6 post dosing
  Adverse events
Incidence of treatment-emergent changes in vital signs in PD patients with multiple ascending doses of anle138b taken 28 days in the non-fasted state (cohort E). | Day 1 to week 6 post dosing
  Blood pressure
Incidence of treatment-emergent changes in vital signs in PD patients with multiple ascending doses of anle138b taken 28 days in the non-fasted state (cohort E). | Day 1 to week 6 post dosing
  Heart rate
Incidence of treatment-emergent changes in vital signs in PD patients with multiple ascending doses of anle138b taken 28 days in the non-fasted state (cohort E). | Day 1 to week 6 post dosing
  Oral temperature
Incidence of treatment-emergent changes in vital signs in PD patients with multiple ascending doses of anle138b taken 28 days in the non-fasted state (cohort E). | Day 1 to week 6 post dosing
  Electrocardiogram (ECG) parameters including QT interval corrected for heart rate using Fridericia's formula (QTcF)
Incidence of treatment-emergent changes in physical examination in PD patients with multiple ascending doses of anle138b taken 28 days in the non-fasted state (cohort E). | Day 1 to week 6 post dosing
  Physical examination findings
Incidence of treatment-emergent changes in clinical laboratory parameters in PD patients with multiple ascending doses of anle138b taken 28 days in the non-fasted state (cohort E). | Day 1 to 24 hours post dosing
  Clinical laboratory Tests: Hematology
Incidence of treatment-emergent changes in clinical laboratory parameters in PD patients with multiple ascending doses of anle138b taken 28 days in the non-fasted state (cohort E). | Day 1 to 24 hours post dosing
  Clinical chemistry: Renal function tests
Incidence of treatment-emergent changes in clinical laboratory parameters in PD patients with multiple ascending doses of anle138b taken 28 days in the non-fasted state (cohort E). | Day 1 to 24 hours post dosing
  Clinical chemistry: Hepatic enzymes
Incidence of treatment-emergent changes in clinical laboratory parameters in PD patients with multiple ascending doses of anle138b taken 28 days in the non-fasted state (cohort E). | Day 1 to 24 hours post dosing
  Clinical chemistry: Electrolytes
Incidence of treatment-emergent changes in clinical laboratory parameters in PD patients with multiple ascending doses of anle138b taken 28 days in the non-fasted state (cohort E). | Day 1 to 24 hours post dosing
  Clinical chemistry: Creatine kinase

SECONDARY OUTCOMES:
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the fasted state (cohorts A-C + D). | Day 1 to day 9
  PK parameter: Tlag for anle138b.
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the fasted state (cohorts A-C + D). | Day 1 to day 9
  PK parameter: Tmax for anle138b.
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the fasted state (cohorts A-C + D). | Day 1 to day 9
  PK parameter: Cmax for anle138b.
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the fasted state (cohort B). | Day 1 to day 9
  PK parameter: C12 for anle138b.
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the fasted state (cohorts A-C + D). | Day 1 to day 9
  PK parameter: C24 for anle138b.
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the fasted state (cohorts A-C + D). | Day 1 to day 9
  PK parameter: AUC(0-tau) for anle138b.
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the fasted state (cohorts A-C + D). | Day 1 to day 9
  PK parameter: Lambda-z for anle138b.
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the fasted state (cohorts A-C + D). | Day 1 to day 9
  PK parameter: T1/2 for anle138b.
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the fasted state (cohorts A-C + D). | Day 1 to day 9
  PK parameter: Accumulation ratio for Cmax (Day 7) for anle138b.
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the fasted state (cohorts A-C + D). | Day 1 to day 9
  PK parameter: Accumulation ratio for AUC (Day 7) for anle138b.
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the fed state (Cohorts A and B). | From fed dosing to 48 hours post dosing.
  PK parameter: Cmax for anle138b.
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the fed state (Cohorts A and B). | From fed dosing to 48 hours post dosing.
  PK parameter: AUC(0-24) for anle138b.
Effect of multiple ascending doses of anle138b on the motor status of PD patients | Admission to follow-up visit (days 14-16 for cohorts A and B; days 12-14 for cohort C; week 6 for cohorts D and E)
  Changes from baseline in the "Movement Disorder Society-sponsored revision of the Unified PD Rating Scale" (MDS-UPDRS) ranging from 0 to 260 points with less points meaning less severity.
Effect of multiple doses of anle138b on the CSF levels of anle138b in PD patients | single time point 3 hours post dose on dosing day 5 (cohort B)
  Quantification of anle138b
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the non-fasted state (cohort E) | Day 1 to day 30
  PK parameter: Tlag for anle138b
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the non-fasted state (cohort E) | Day 1 to day 30
  PK parameter: Tmax for anle138b
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the non-fasted state (cohort E) | Day 1 to day 30
  PK parameter: Cmax for anle138b
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the non-fasted state (cohort E) | Day 1 to day 30
  PK parameter: C12 for anle138b
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the non-fasted state (cohort E) | Day 1 to day 30
  PK parameter: C24 for anle138b
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the non-fasted state (cohort E) | Day 1 to day 30
  PK parameter: AUC(0-tau) for anle138b
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the non-fasted state (cohort E) | Day 1 to day 30
  PK parameter: Lambda-z for anle138b
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the non-fasted state (cohort E) | Day 1 to day 30
  PK parameter: T1/2 for anle138b
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the non-fasted state (cohort E) | Day 1 to day 30
  PK parameter: Accumulation ratio for Cmax for anle138b
Oral pharmacokinetics (PK) of multiple ascending doses of anle138b in PD patients taken in the non-fasted state (cohort E) | Day 1 to day 30
  PK parameter: Accumulation ratio for AUC for anle138b

CONTACTS AND LOCATIONS:
Overall Officials: Nand Singh, BSc, MD, DPM, MFPM, Principal Investigator — Quotient Sciences Mere Way Ruddington Fields Ruddington Nottingham NG11 6JS, UK; Jonathan Evans, MD, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagner J, Ryazanov S, Leonov A, Levin J, Shi S, Schmidt F, Prix C, Pan-Montojo F, Bertsch U, Mitteregger-Kretzschmar G, Geissen M, Eiden M, Leidel F, Hirschberger T, Deeg AA, Krauth JJ, Zinth W, Tavan P, Pilger J, Zweckstetter M, Frank T, Bahr M, Weishaupt JH, Uhr M, Urlaub H, Teichmann U, Samwer M, Botzel K, Groschup M, Kretzschmar H, Griesinger C, Giese A. Anle138b: a novel oligomer modulator for disease-modifying therapy of neurodegenerative diseases such as prion and Parkinson's disease. Acta Neuropathol. 2013 Jun;125(6):795-813. doi: 10.1007/s00401-013-1114-9. Epub 2013 Apr 19. PMID 23604588
- [Background] Levin J, Schmidt F, Boehm C, Prix C, Botzel K, Ryazanov S, Leonov A, Griesinger C, Giese A. The oligomer modulator anle138b inhibits disease progression in a Parkinson mouse model even with treatment started after disease onset. Acta Neuropathol. 2014 May;127(5):779-80. doi: 10.1007/s00401-014-1265-3. Epub 2014 Mar 11. No abstract available. PMID 24615514
- [Background] Heras-Garvin A, Weckbecker D, Ryazanov S, Leonov A, Griesinger C, Giese A, Wenning GK, Stefanova N. Anle138b modulates alpha-synuclein oligomerization and prevents motor decline and neurodegeneration in a mouse model of multiple system atrophy. Mov Disord. 2019 Feb;34(2):255-263. doi: 10.1002/mds.27562. Epub 2018 Nov 19. PMID 30452793
- [Background] Wegrzynowicz M, Bar-On D, Calo' L, Anichtchik O, Iovino M, Xia J, Ryazanov S, Leonov A, Giese A, Dalley JW, Griesinger C, Ashery U, Spillantini MG. Depopulation of dense alpha-synuclein aggregates is associated with rescue of dopamine neuron dysfunction and death in a new Parkinson's disease model. Acta Neuropathol. 2019 Oct;138(4):575-595. doi: 10.1007/s00401-019-02023-x. Epub 2019 May 31. PMID 31165254
- [Background] Wagner J, Krauss S, Shi S, Ryazanov S, Steffen J, Miklitz C, Leonov A, Kleinknecht A, Goricke B, Weishaupt JH, Weckbecker D, Reiner AM, Zinth W, Levin J, Ehninger D, Remy S, Kretzschmar HA, Griesinger C, Giese A, Fuhrmann M. Reducing tau aggregates with anle138b delays disease progression in a mouse model of tauopathies. Acta Neuropathol. 2015 Nov;130(5):619-31. doi: 10.1007/s00401-015-1483-3. Epub 2015 Oct 6. PMID 26439832
- [Background] Martinez Hernandez A, Urbanke H, Gillman AL, Lee J, Ryazanov S, Agbemenyah HY, Benito E, Jain G, Kaurani L, Grigorian G, Leonov A, Rezaei-Ghaleh N, Wilken P, Arce FT, Wagner J, Fuhrmann M, Caruana M, Camilleri A, Vassallo N, Zweckstetter M, Benz R, Giese A, Schneider A, Korte M, Lal R, Griesinger C, Eichele G, Fischer A. The diphenylpyrazole compound anle138b blocks Abeta channels and rescues disease phenotypes in a mouse model for amyloid pathology. EMBO Mol Med. 2018 Jan;10(1):32-47. doi: 10.15252/emmm.201707825. PMID 29208638
- See also: Sponsor Homepage — http://www.modag.net